CLINICAL TRIAL: NCT04159038
Title: Integrating WIC With Early Childhood Systems of Developmental Care
Acronym: CDC-WIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study sites were closed in March 2020, due to COVID-19 and did not re-open; follow-up data were collected for 6 months subsequently of already enrolled subjects
Sponsor: Oregon Health and Science University (Other)
Collaborators: Oregon WIC Program (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Katharine Zuckerman, MD MPH, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY00019833; 19-3773 PO# 2000043062 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Developmental Disability; Food Assistance; Health Care Disparity
Keywords: Pilot Projects; Randomized Controlled Trial
MeSH Terms: conditions — Developmental Disabilities | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parents in the immediate intervention arm sign a study consent that is integrated into the Women, Infants, & Children (WIC) Referral Form. They also complete a brief demographic survey. No consent is necessary in the delayed intervention arm as only aggregate information will be reported to the study team by Early Intervention/Early Childhood Special Education. EI/ECSE referrals are tracked from clinics in both arms for 6 months in ecWeb. At the end of the data collection period, the study team will meet to refine the intervention based on the experience with the immediate intervention group. Qualitative Interviews will take place with WIC staff, parents who indicate interest, EI/ECSE staff, and primary care providers during and after the post-intervention data collection period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): Parents in the immediate intervention arm sign a study consent that is integrated into the WIC Referral Form. They also complete a brief demographic survey. No consent is necessary in the delayed intervention arm as only aggregate information will be reported to the study team by EI/ECSE. EI/ECSE referrals are tracked from clinics in both arms for 6 months in ecWeb. At the end of the data collection period, the study team will meet to refine the intervention based on the experience with the immediate intervention group. Qualitative Interviews will take place with WIC staff, parents who indicate interest, EI/ECSE staff, and primary care providers during and after the post-intervention data collection period.
  Interventions: Other: Intervention Group
- Delayed Intervention Group (Other): 6 months after the immediate intervention group receives their training, the delayed intervention group will receive the training. Prior to implementation of the training in the delayed intervention group, the study team will meet with the Stakeholder Advisory Board. It will review interim results and consider the efficacy of the intervention as a whole. Based on actual use patterns and stakeholder feedback, the investigators will make improvements to the intervention prior to implementing it in the delayed intervention group.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Intervention Group — The immediate intervention group will receive training on how to identify children at risk for developmental disabilities and how to refer to Early Intervention/Early Childhood Special Education.
  Arms: Immediate Intervention Group
Other: Control group — The control group will continue usual WIC care.
  Arms: Delayed Intervention Group

SUMMARY:
This study's goals are to improve connections between Oregon Women, Infants, & Children (WIC) clinics, primary care providers, and Early Intervention/Early Childhood Special Education programs (EI/ECSE), in order to help children with suspected developmental delays get the services they need.

DETAILED DESCRIPTION:
Disparities exist in early identification of developmental disabilities, particularly for families from low-income and/or racial ethnic minority backgrounds. As WIC has frequent contact with children and families in the first five years of life, it is optimally positioned to play a unique role in early identification of developmental disabilities. However, WIC staff are not formally trained in child development outside of program's primary focus on nutrition and supporting the feeding relationship nor is formal screening for potential developmental delays an allowable WIC expense. In our prior research Oregon WIC staff reported being frequently asked by parents about potential concerns yet they also reported not being well connected to pediatric primary care, Part C Early Intervention (EI), or other resources who could further assess these concerns. In this study the investigators propose to design and pilot test a 2-part intervention to enhance the link between WIC and early childhood resources. The 2-part intervention includes: (1) WIC staff training delivered at the Local Agency which will: build staff confidence in discussing developmental concerns with families, familiarize staff with the CDC Learn the Signs Act Early (LTSAE) material which may be used to support those conversations, provide easy tips for encouraging early language and literacy development with parents, and study procedures (2) the creation of a standardized, direct, closed-loop referral process from WIC to EI for families with an identified concern who agree to the referral. EI will notify the child's primary care provider of the referral as per usual EI protocol. A referral form has been approved by the Oregon Department of Education (ODE) to support the direct referral from WIC to EI, meeting all ODE FERPA requirements. In addition, a data use agreement has been approved by ODE to allow the study team to access data on referred children to determine if they completed further assessment and the given diagnosis (if any). While our primary quantitative outcomes of interest are the number of children with a potential developmental concern who are referred directly from WIC to EI, the timing of follow-up assessment by EI from that referral, services plan & start of services; the project really centers on improving processes between organizations who are key stakeholders in referral, assessment, and treatment. Therefore, secondary outcomes include feasibility and acceptability of the intervention amongst WIC staff, EI staff and primary care providers Upon completion of the study the investigators hope to apply our findings to scale up the WIC staff training and closed-loop referral process to take it Statewide. If successful the investigators will disseminate findings through the National WIC Association to encourage other State and Tribal WIC Authorities to adopt our procedures as best practices.

ELIGIBILITY:
Inclusion Criteria:

* The primary subject population of interest are Women, Infants, & Children families who in the course of a WIC visit identify a potential developmental concern and agree to a direct referral from WIC to Early Intervention to further assess that concern. To be eligible for the study, the parent/guardian must speak English or Spanish. The child with the identified concern must be under 54 months of age as the investigators will need to follow the child for 6 months to determine initial outcomes and children are no longer eligible for WIC after their 5th birthday.

WIC staff at the 4 intervention agencies, EI staff in the 4 communities in which the 4 intervention WIC Local Agencies are located, and primary care providers (PCPs) who have had a patient referred to EI directly from WIC will all be invited to participate in a telephone interview to give their perspective on the process. The only staff inclusion requirement is that these staff are currently working in their professional role in the county studied.

Exclusion Criteria:

* Family speaks language that isn't English or Spanish. Child is older than 54 months.

Staff does not work in their professional role in the county studied.

Max Age: 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2020-01-10 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
% of Women, Infants, & Children (WIC) participant visits with Early Intervention/Early Childhood Special Education (EI/ECSE) referral. | Start of intervention for 6 months
  in immediate versus delayed intervention arms, to understand if the intervention boosted EI/ECSE referral rates.
% EI/ECSE referrals evaluated by EI/ECSE | Start of intervention for 6 months
  by 6 months after referral, in both arms, to see if increased referral actually results in increased EI/ECSE evaluation.
Time from referral to evaluation | Start of intervention for 6 months
  in both arms, to see if the intervention accelerated EI/ECSE evaluation.

SECONDARY OUTCOMES:
% of those found eligible on EI/ECSE treatment, 6-months post referral | Start of intervention for 6 months
  to see if the intervention increased the number of children receiving treatment services in EI/ECSE.
% of public-health identified children referred to EI/ECSE by WIC | Start of intervention for 6 months
  to see if WIC can identify and refer children who are high-risk but not otherwise accessing developmental care.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine Zuckerman, M.D., M.P.H., Principal Investigator — Oregon Health and Science University
Locations (4):
- United States (4):
  - Deschutes County WIC, Bend, Oregon
  - Josephine County WIC, Grants Pass, Oregon
  - Washington County WIC, Hillsboro, Oregon
  - Jefferson County WIC, Madras, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Disability Research and Dissemination Center- Grants Awarded through the DRDC Mechanism — https://www.disabilityresearchcenter.com/research/awarded-grants/